CLINICAL TRIAL: NCT04030351
Title: Effect of Dried Fruit Intake on Acid-base Balance in Community Dwelling Adults
Brief Title: Effect of Dried Fruit Intake on Acid-base Balance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Institution shut down due to COVID-19
Sponsor: Tufts University (Other)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Director of Bone Metabolism Laboratory, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2980
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Acid-Base Balance Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dried fruit (Experimental): 100 g per day of dried fruit
  Interventions: Other: food - dried fruit
- no dried fruit (No Intervention): no intervention to be given

INTERVENTIONS:
Other: food - dried fruit — raisins, apricots, figs, and pineapple
  Arms: dried fruit

SUMMARY:
Most adults consume acid-producing diets because their high intake of protein and/or cereal grains in relation to their intake of fruits and vegetables. This study is being done to determine whether acid-base balance can be restored by the addition of dried fruits to the diet. In this study adults with low usual fruit intake will be provided with either 100 g per day of a mix of dried fruits or no dried fruit. Participants will be followed for 1 year. Acid-base status will be assessed by measuring the acid content in 24-hour urine collections.

DETAILED DESCRIPTION:
Most adults consume acid-producing diets because their intake of protein and/or cereal grains is high in relation to their intake of fruits and vegetables. Supplementation with alkaline salts such as potassium bicarbonate and potassium citrate have been shown to reduce 24-hr urinary net acid excretion (NAE) in healthy adults. This approach requires taking many capsules daily, in split doses after each meal with a full glass of water. An alternative and perhaps more acceptable approach to achieving acid-base balance for most adults may be to modify their diet by increasing intake of alkali-producing foods, such as fruit. Maintaining acid base balance may be important for preserving bone and muscle and renal function and other outcomes but this has not been established. The investigators propose to determine whether adults who are provided with 100 g per day of a selection of dried fruits will actually consume enough of it to correct their acid-producing diets, as evidenced by a lowering of their urinary NAE. The investigators will also determine whether and how participants will alter their overall diets or their body weight when provided with the dried fruit. The comparator group will receive no dried fruit (or other intervention).

ELIGIBILITY:
Inclusion Criteria:

* usual self-reported fruit intake not greater than 2.5 servings per day
* adequate dentition to chew dried fruit
* willing to avoid potassium supplements during the study
* willing to avoid antacids other than Pepto Bismol during the study

Exclusion Criteria:

Conditions

* diabetes or fasting plasma glucose on screening >125 mg/dl
* untreated thyroid disease
* untreated parathyroid disease
* cirrhosis
* unstable heart disease
* osteoporosis of the spine or hip
* alcohol use > 2 drinks per day
* chronic diarrheal syndrome
* estimated glomerular filtration rate < 50 ml/min
* serum potassium >5.3 meq/L
* abnormal serum calcium
* dysphasia
* malabsorption
* inflammatory bowel disease
* celiac disease
* chronic constipation
* gastric bypass surgery
* non-English speaking Medications
* potassium sparing diuretics
* oral glucocorticoids
* immunosuppressant drugs
* anabolic steroids in last 6 months
* estrogen in last 6 months
* osteoporosis treatment in the last 12 months with teriparatide abaloparatide calcitonin raloxifene denosumab
* osteoporosis treatment with a bisphosphonate in the last 2 years
* regular use of antacids > 3 times per week
* regular use of laxatives > 3 times per week
* any medication taken to alter appetite

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
change in 24-hour urinary NAE | 12 month
  NAE reflects net acid-base balance

SECONDARY OUTCOMES:
rate of adherence with dried fruit | 12 months
  weight of dispensed fruit consumed, calculated as weight of fruit dispensed minus the weight of fruit returned
change in 24-hour urinary N-telopeptide | 12 months
  a measure of bone resorption
change in fat to lean tissue mass ratio | 12 months
  a measure of change in body composition by dual-energy x-ray absorptiometry (DXA:)
change in bone mineral density at the total body | 12 months
  measured by DXA
change in body weight | 12 months
  measured on a standard scale
change in grip strength | 12 months
  hand grip strength in kilograms assessed by a hand held dynamometer
Mediterranean diet score | 12 months
  a 14-item scale of adherence to a healthy Mediterranean style diet; a higher score represents a better diet
change in bone mineral density of the spine | 12 months
  measured by DXA
change in bone mineral density of the hip | 12 months
  measured by DXA
Health Aging and Body Composition-leg strength | 12 months
  defined as ability to do 5 repeated chair stands; assessed on a 4-point scale; a higher score represents a better performance
Health Aging and Body Composition - standing balance | 12 months
  defined as ability to stand in tandem position measured on a 4-point scale; a higher score represents a better performance
Health Aging and Body Composition- gait speed | 12 months
  defined as usual gait speed of performing a 6-meter walk; assessed on a 4-point scale; a higher score represents a better performance
Health Aging and Body Composition-physical performance battery | 12 months
  The total score is 12 points, representing the sum of the 4-point scores of the 3 domains (strength, balance and gait speed). A higher score represents a better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No